CLINICAL TRIAL: NCT05215054
Title: Clinical Study for the Safety and Effectiveness of Use of an Injectable Medical Device GANA V® for Facial Aesthetic Treatment
Brief Title: Clinical Study for the Evaluation of the Safety and Effectiveness of Use of a Poly-L Lactic Acid Injectable Filler for the Aesthetic Treatment of Nasolabial Folds
Acronym: PLLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Co., Ltd (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E0787; 2021-A02451-40 (Other: ANSM)
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Wrinkle

STUDY DESIGN:
Intervention Model Description: All participants will receive both fillers
Masking Description: Participants and investigators assessors will not know which filler was used on each side of the face (hemi-face design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gana V versus Sculptra (Experimental): Participants will receive both Gana V and Sculptra: one in each nasolabial folds
  Interventions: Device: Gana V®; Device: Sculptra®

INTERVENTIONS:
Device: Gana V® — Injection in the deep dermis and subcutaneous layer of the nasolabial fold on D0 (initial injection) and 1 month and a half after initial injection if necessary (optional touch-up).
Device: Sculptra® — Injection in the deep dermis and subcutaneous layer of the nasolabial fold on D0 (initial injection) and 1 month and a half after initial injection if necessary (optional touch-up).

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of Gana V, a Poly L-lactic acid filler for the aesthetic treatment of nasolabial folds, in comparison with Sculptra.

DETAILED DESCRIPTION:
A screening visit will allow to inform and preselect the participants.

On D0, baseline scoring, fringe projection acquisitions and photographs will be done before injection. Eligible participants will receive a first injection of the two products according to the randomization list. Immediately after injection, injector's treatment satisfaction will be collected. Investigator evaluator will collect Adverse Events (AEs) and Injection Site Reactions (ISRs) immediately after injection.

A month and a half after initial injection (M11/2), clinical scoring, fringe projection acquisitions and photographs will be done before touch-up (if applicable). Participant's treatment satisfaction and injector's treatment satisfaction (if applicable) will be collected. A touch-up injection will be made if necessary, according to injector and participant opinion. Investigator evaluator will collect AEs and ISRs before and after touch-up if applicable.

Three (M3), six (M6), nine (M9), twelve (M12), eighteen (M18) and twenty-four (M24) months after initial injection, clinical scoring, fringe projection acquisitions and photographs will be done. Participant's treatment satisfaction will be collected. Investigator evaluator will collect AEs and ISRs

ELIGIBILITY:
Inclusion Criteria:

* Subject with moderate to severe nasolabial folds as determined by a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 on both folds at the pre-treatment evaluation.
* Subject wiling to abstain from other facial procedures (i.e., dermal fillers, toxin treatments, laser, microdermal abrasion, chemical peels, non-invasive skin-tightening) during the whole study period.
* Subject, psychologically able to understand the study related information and to give a written informed consent.
* Subject having given freely and expressly his/her informed consent.
* Subject willing to have photographs of the face taken.
* Subject affiliated to a health social security system.
* Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit and during the whole study period.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject with a scar, moles, pigment disorders or anything on the face which might interfere with the evaluation.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment
* Subject participation to another research on human beings or who is in an exclusion period of one.
* Subject having received 4500 euros indemnities for participation in research involving human beings in the 12 previous months, including participation in the present study.
* Subject suspected to be non-compliant according to the investigator's judgment.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (e.g. acne, mycosis, papilloma, chronic eczema, atopic dermatitis…). Subject with labial herpes in the last 2 years is not eligible even if asymptomatic at time of screening visit.
* Subject with an abscess, unhealed wound, or a cancerous or precancerous lesion on the studied zone.
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Subject with a tendency to develop keloids or hypertrophic scarring.
* Subject having history of allergy or anaphylactic shock including hypersensitivity to Poly-l-lactic acid, to lidocaine or to one of the components of the tested devices or antiseptic solution.
* Subject having received treatment with a laser, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to screening visit.
* Subject having received injection with a resorbable filling product in the face area within the past 12 months prior to screening visit.
* Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …) on the face.
* Subject having received at any time a treatment with tensor threads on the face.
* Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.
* Subject using medication such as aspirin, nonsteroidal anti-inflammatory drugs (NSAID) (ibuprofen, naproxen, …), antiplatelet agents, anticoagulants or other substances known to prolong bleeding time within 1 week prior to injection visits.
* Subject undergoing a topical treatment on the test area or a systemic treatment:

  * Antihistamines during the 2 weeks prior to screening visit.
  * Immunosuppressors and/or corticoids during the 4 weeks prior to screening visit.
  * Retinoids during the 6 months prior to screening visit.
* Intensive exposure to sunlight or UV-rays within the previous month before and after injection visits.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Morel, Doctor, Principal Investigator — Eurofins Dermscan Pharmascan
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Kim HJ, Han WY, Yon DK. Final Report on the Safety and Efficacy of Poly-L-Lactic Acid Filler (Gana V) Injection for the Correction of Nasolabial Fold: A Double-Blind, Non-Inferiority, Randomized, Split-Face Controlled Trial. Aesthetic Plast Surg. 2025 Sep 2. doi: 10.1007/s00266-025-05190-3. Online ahead of print. PMID 40897963
- [Derived] Han WY, Kim HJ, Kwon R, Kang SM, Yon DK. Safety and Efficacy of Poly-L-Lactic Acid Filler (Gana V vs. Sculptra) Injection for Correction of the Nasolabial Fold: A Double-Blind, Non-Inferiority, Randomized, Split-Face Controlled Trial. Aesthetic Plast Surg. 2023 Oct;47(5):1796-1805. doi: 10.1007/s00266-023-03600-y. Epub 2023 Aug 25. PMID 37626137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation was initiated on 7 March 2022 (first subject first visit). Subjects were recruited from one investigational center, Eurofins Dermscan Pharmascan centre in Villeurbanne, France.The last subject was screened on 4 May 2022, and the recruitment period lasted 58 days.
Pre-assignment Details: 4 subjects were enrolled but not randomized in the study due to consent withdrawal or because they were lost to follow-up
Units Other Than Participants: Nasolabial fold
Groups:
- Gana V: Participants received Gana V in one nasolabial fold (as per randomization list-split face design).1ml maximum of product could be used at the initial visit (D0) and 1ml maximum could be used 1 month and a half after the initial visit (touch-up not mandatory).
- Sculptra: Participants received Sculptra in the other nasolabial fold (as per randomization list-split face design). 1ml maximum of product could be used at the initial visit (D0) and 1ml maximum could be used 1 month and a half after the initial visit (touch-up not mandatory).
Period: Overall Study
Arm/Group | Gana V | Sculptra
Started | 55; 55 Nasolabial fold | 55; 55 Nasolabial fold
Completed | 49; 49 Nasolabial fold | 49; 49 Nasolabial fold
Not Completed | 6; 6 Nasolabial fold | 6; 6 Nasolabial fold
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Gana V Versus Sculptra: Participants received both Gana V and Sculptra: one in each nasolabial folds
Arm/Group | Gana V Versus Sculptra
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Nasolabial Folds Severity Score on the Wrinkle Severity Rating Scale (WSRS) 6 Months After Treatment
Description: The Wrinkle Severity Rating Scale is a scale for measurement of the nasolabial folds wrinkles severity.
  The scale ranges from Grade 1 (absent-better outcome) to Grade 5 (extreme-worse outcome) Change of grades was calculated as the value at 6 months minus the value at baseline. To observe an improvement of the nasolabial folds wrinkles, a decrease of the mean score was expected.
Time Frame: Baseline and Month 6
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Nasolabial fold
Groups:
- Sculptra: Participants received Sculptra in one nasolabial fold (as per randomization list-split face design).1ml maximum of product could be used at the initial visit (D0) and 1ml maximum could be used 1 month and a half after the initial visit (touch-up not mandatory).
- Gana V Versus Sculptra: Comparison between results obtained for Gana V and results obtained for Sculptra
Arm/Group | Gana V | Sculptra | Gana V Versus Sculptra
Number analyzed (Participants) | 53 | 53 | 53
Number analyzed (Nasolabial fold) | 53 | 53 | 106
score on a scale | -0.3 [-0.4 to -0.1] | -0.2 [-0.3 to -0.1] | -0.1 [-0.2 to 0.1]
Statistical Analysis 1: Comparison: Gana V vs Sculptra; Difference of changes from baseline in WSRS score for Gana V versus Sculptra; Test type: Non-Inferiority — Non-inferiority will be demonstrated if the upper limit of the two-sided 95%CI of the difference of changes from baseline between test device and control is inferior or equal to 0.5; Non-inferiority will be demonstrated if the upper limit of the two-sided 95%CI of the difference of changes from baseline between test device and control is inferior or equal to 0.5.To assess assay sensitivity, the proportion of responders with Gana V®, defined as improvement of ≥1-grade in the WSRS when compared to D0 pre-injection must be ≥50% at the 6 months visit after baseline

2. Secondary Outcome: Change From Baseline in the Nasolabial Folds Severity Score on the Wrinkle Severity Rating Scale (WSRS)
Description: The Wrinkle Severity Rating Scale is a scale for measurement of the nasolabial folds wrinkles severity.
  The scale ranges from Grade 1 (absent-better outcome) to Grade 5 (extreme-worse outcome) Change of grades was calculated as the value at month X minus the value at baseline. To observe an improvement of the nasolabial folds wrinkles, a decrease of the mean score was expected.
Time Frame: Baseline, Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Nasolabial fold
Groups:
- Gana V Versus Sculptra: All participants
- Gana V: All nasolabial fold who received injection with Gana V®
- Sculptra: All nasolabial fold who received injection with Sculptra®
Arm/Group | Gana V Versus Sculptra | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55 | 55
Number analyzed (Nasolabial fold) | 110 | 55 | 55
score on a scale
  Change from baseline (D0 visit) to M11/2 visit | -0.1 (0.3) | -0.1 (0.3) | -0.0 (0.2)
  Change from baseline (D0 visit) to M3 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M3 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M3 visit | 0.0 (0.2) | -0.1 (0.3) | -0.1 (0.3)
  Change from baseline (D0 visit) to M6 visit: number analyzed (Participants) | 53 | 53 | 53
  Change from baseline (D0 visit) to M6 visit: number analyzed (Nasolabial fold) | 106 | 53 | 53
  Change from baseline (D0 visit) to M6 visit | -0.1 (0.5) | -0.3 (0.4) | -0.2 (0.4)
  Change from baseline (D0 0visit) to M9 visit: number analyzed (Participants) | 48 | 48 | 48
  Change from baseline (D0 0visit) to M9 visit: number analyzed (Nasolabial fold) | 96 | 48 | 48
  Change from baseline (D0 0visit) to M9 visit | -0.2 (0.6) | -0.4 (0.5) | -0.3 (0.4)
  Change from baseline (D0 visit) to M12 visit: number analyzed (Participants) | 47 | 47 | 47
  Change from baseline (D0 visit) to M12 visit: number analyzed (Nasolabial fold) | 94 | 47 | 47
  Change from baseline (D0 visit) to M12 visit | -0.1 (0.5) | -0.4 (0.6) | -0.3 (0.5)
  Change from baseline (D0 visit) to M18 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M18 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M18 visit | -0.1 (0.3) | -0.3 (0.5) | -0.2 (0.5)
  Change from baseline (D0 visit) to M24 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M24 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M24 visit | -0.1 (0.3) | -0.2 (0.5) | -0.1 (0.4)

3. Secondary Outcome: WSRS Responders Rate
Description: The Wrinkle Severity Rating Scale is a scale for measurement of the nasolabial folds wrinkles severity.
  The scale ranges from Grade 1 (absent-better outcome) to Grade 5 (extreme-worse outcome) Responders rate = percentage of participants with an improvement of at least one grade in WSRS compared to baseline score. An improvement represents a decrease in WSRS (from grade 5 to grade 4 for instance)
Time Frame: Baseline, Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value.
Measure: Count of Participants; unit: Participants
Arm/Group | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55
Participants
  Responder rate from baseline (D0 visit) to M11/2 visit: Responder | 5 | 2
  Responder rate from baseline (D0 visit) to M11/2 visit: Not responder | 50 | 53
  Responder rate from baseline (D0 visit) to M3 visit: number analyzed (Participants) | 49 | 49
  Responder rate from baseline (D0 visit) to M3 visit: Responder | 6 | 6
  Responder rate from baseline (D0 visit) to M3 visit: Not responder | 43 | 43
  Responder rate from baseline (D0 visit) to M6 visit: number analyzed (Participants) | 53 | 53
  Responder rate from baseline (D0 visit) to M6 visit: Responder | 14 | 11
  Responder rate from baseline (D0 visit) to M6 visit: Not responder | 39 | 42
  Responder rate from baseline (D0 visit) to M9 visit: number analyzed (Participants) | 48 | 48
  Responder rate from baseline (D0 visit) to M9 visit: Responder | 20 | 13
  Responder rate from baseline (D0 visit) to M9 visit: Not responder | 28 | 35
  Responder rate from baseline (D0 visit) to M12 visit: number analyzed (Participants) | 47 | 47
  Responder rate from baseline (D0 visit) to M12 visit: Responder | 16 | 13
  Responder rate from baseline (D0 visit) to M12 visit: Not responder | 31 | 34
  Responder rate from baseline (D0 visit) to M18 visit: number analyzed (Participants) | 49 | 49
  Responder rate from baseline (D0 visit) to M18 visit: Responder | 12 | 9
  Responder rate from baseline (D0 visit) to M18 visit: Not responder | 37 | 40
  Responder rate from baseline (D0 visit) to M24 visit: number analyzed (Participants) | 49 | 49
  Responder rate from baseline (D0 visit) to M24 visit: Responder | 10 | 6
  Responder rate from baseline (D0 visit) to M24 visit: Not responder | 39 | 43

4. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Responder Rate
Description: Percentage of participants with an improvement on GAIS. A responder is defined as a subject having "Improved", "Much improved" or "Very much improved" score according to GAIS.
Time Frame: Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value.
Measure: Count of Participants; unit: Participants
Arm/Group | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55
Participants
  Evaluated by the independent blind evaluator at M11/2: Responder | 20 | 18
  Evaluated by the independent blind evaluator at M11/2: Not responder | 35 | 37
  Evaluated by the independent blind evaluator at M3: number analyzed (Participants) | 49 | 49
  Evaluated by the independent blind evaluator at M3: Responder | 21 | 17
  Evaluated by the independent blind evaluator at M3: Not responder | 28 | 32
  Evaluated by the independent blind evaluator at M6: number analyzed (Participants) | 53 | 53
  Evaluated by the independent blind evaluator at M6: Responder | 38 | 29
  Evaluated by the independent blind evaluator at M6: Not responder | 15 | 24
  Evaluated by the independent blind evaluator at M9: number analyzed (Participants) | 48 | 48
  Evaluated by the independent blind evaluator at M9: Responder | 32 | 31
  Evaluated by the independent blind evaluator at M9: Not responder | 16 | 17
  Evaluated by the independent blind evaluator at M12: number analyzed (Participants) | 46 | 46
  Evaluated by the independent blind evaluator at M12: Responder | 30 | 28
  Evaluated by the independent blind evaluator at M12: Not responder | 16 | 18
  Evaluated by the independent blind evaluator at M18: number analyzed (Participants) | 49 | 49
  Evaluated by the independent blind evaluator at M18: Responder | 26 | 27
  Evaluated by the independent blind evaluator at M18: Not responder | 23 | 22
  Evaluated by the independent blind evaluator at M24: number analyzed (Participants) | 49 | 49
  Evaluated by the independent blind evaluator at M24: Responder | 16 | 17
  Evaluated by the independent blind evaluator at M24: Not responder | 33 | 32
  Evaluated by the subjects at M11/2: Responder | 27 | 27
  Evaluated by the subjects at M11/2: Not responder | 28 | 28
  Evaluated by the subjects at M3: number analyzed (Participants) | 53 | 53
  Evaluated by the subjects at M3: Responder | 34 | 32
  Evaluated by the subjects at M3: Not responder | 19 | 21
  Evaluated by the subjects at M6: number analyzed (Participants) | 53 | 53
  Evaluated by the subjects at M6: Responder | 35 | 34
  Evaluated by the subjects at M6: Not responder | 18 | 19
  Evaluated by the subjects at M9: number analyzed (Participants) | 47 | 48
  Evaluated by the subjects at M9: Responder | 32 | 28
  Evaluated by the subjects at M9: Not responder | 15 | 20
  Evaluated by the subjects at M12: number analyzed (Participants) | 47 | 47
  Evaluated by the subjects at M12: Responder | 29 | 28
  Evaluated by the subjects at M12: Not responder | 18 | 19
  Evaluated by the subjects at M18: number analyzed (Participants) | 49 | 49
  Evaluated by the subjects at M18: Responder | 29 | 31
  Evaluated by the subjects at M18: Not responder | 20 | 18
  Evaluated by the subjects at M24: number analyzed (Participants) | 49 | 49
  Evaluated by the subjects at M24: Responder | 21 | 24
  Evaluated by the subjects at M24: Not responder | 28 | 25

5. Secondary Outcome: Change From Baseline in Nasolabial Folds Average Depth (mm)
Description: The average depth of the nasolabial folds wrinkles was calculated using a fringe projection system. An increase of the mean value means a positive outcome.
  Change was calculated as the value at each follow-up visit minus the value at baseline
Time Frame: Baseline, Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Nasolabial fold
Arm/Group | Gana V Versus Sculptra | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55 | 55
Number analyzed (Nasolabial fold) | 110 | 55 | 55
mm
  Change from baseline (D0 visit) to M11/2 visit | 0.004 (0.019) | 0.018 (0.017) | 0.014 (0.016)
  Change from baseline (D0 visit) to M3 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M3 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M3 visit | 0.008 (0.022) | 0.029 (0.025) | 0.021 (0.017)
  Change from baseline (D0 visit) to M6 visit: number analyzed (Participants) | 51 | 51 | 51
  Change from baseline (D0 visit) to M6 visit: number analyzed (Nasolabial fold) | 102 | 51 | 51
  Change from baseline (D0 visit) to M6 visit | 0.005 (0.026) | 0.029 (0.028) | 0.024 (0.021)
  Change from baseline (D0 visit) to M9 visit: number analyzed (Participants) | 48 | 48 | 48
  Change from baseline (D0 visit) to M9 visit: number analyzed (Nasolabial fold) | 96 | 48 | 48
  Change from baseline (D0 visit) to M9 visit | 0.008 (0.024) | 0.031 (0.028) | 0.023 (0.021)
  Change from baseline (D0 visit) to M12 visit: number analyzed (Participants) | 46 | 46 | 46
  Change from baseline (D0 visit) to M12 visit: number analyzed (Nasolabial fold) | 92 | 46 | 46
  Change from baseline (D0 visit) to M12 visit | 0.008 (0.027) | 0.029 (0.030) | 0.021 (0.020)
  Change from baseline (D0 visit) to M18 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M18 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M18 visit | 0.008 (0.034) | 0.029 (0.027) | 0.020 (0.027)
  Change from baseline (D0 visit) to M24 visit: number analyzed (Participants) | 46 | 46 | 47
  Change from baseline (D0 visit) to M24 visit: number analyzed (Nasolabial fold) | 92 | 46 | 47
  Change from baseline (D0 visit) to M24 visit | -0.002 (0.033) | 0.016 (0.022) | 0.016 (0.031)

6. Secondary Outcome: Change From Baseline in Nasolabial Folds Volume
Description: The volume of the nasolabial folds wrinkles was calculated using a fringe projection system. A decrease of the volume means a positive outcome.
Time Frame: Baseline, Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value
Measure: Mean (Standard Deviation); unit: mm3
Units Other Than Participants: Nasolabial fold
Arm/Group | Gana V Versus Sculptra | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55 | 55
Number analyzed (Nasolabial fold) | 110 | 55 | 55
mm3
  Change from baseline (D0 visit) to M11/2 visit | -0.606 (1.707) | -1.444 (1.692) | -0.838 (1.408)
  Change from baseline (D0 visit) to M3 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M3 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M3 visit | -0.840 (1.914) | -2.458 (2.271) | -1.619 (1.938)
  Change from baseline (D0 visit) to M6 visit: number analyzed (Participants) | 51 | 51 | 51
  Change from baseline (D0 visit) to M6 visit: number analyzed (Nasolabial fold) | 102 | 51 | 51
  Change from baseline (D0 visit) to M6 visit | -0.782 (1.918) | -2.591 (2.038) | -1.809 (1.709)
  Change from baseline (D0 visit) to M9 visit: number analyzed (Participants) | 48 | 48 | 48
  Change from baseline (D0 visit) to M9 visit: number analyzed (Nasolabial fold) | 96 | 48 | 48
  Change from baseline (D0 visit) to M9 visit | -1.041 (1.919) | -2.719 (2.059) | -1.677 (1.956)
  Change from baseline (D0 visit) to M12 visit: number analyzed (Participants) | 46 | 46 | 46
  Change from baseline (D0 visit) to M12 visit: number analyzed (Nasolabial fold) | 92 | 46 | 46
  Change from baseline (D0 visit) to M12 visit | -0.832 (1.985) | -2.281 (2.232) | -1.449 (1.707)
  Change from baseline (D0 visit) to M18 visit: number analyzed (Participants) | 49 | 49 | 49
  Change from baseline (D0 visit) to M18 visit: number analyzed (Nasolabial fold) | 98 | 49 | 49
  Change from baseline (D0 visit) to M18 visit | -0.909 (2.383) | -2.351 (2.305) | -1.442 (2.162)
  Change from baseline (D0 visit) to M24 visit: number analyzed (Participants) | 46 | 46 | 47
  Change from baseline (D0 visit) to M24 visit: number analyzed (Nasolabial fold) | 92 | 46 | 47
  Change from baseline (D0 visit) to M24 visit | 0.161 (2.392) | -0.949 (2.031) | -0.939 (2.496)

7. Secondary Outcome: Proportion of Satisfied Participants
Description: Percentage of participants with positive answers to an internal questionnaire
Time Frame: Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value
Measure: Count of Participants; unit: Participants
Arm/Group | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55
Participants
  Are you satisfied with how your nasolabial fold looks? at M11/2: Satisfied | 28 | 29
  Are you satisfied with how your nasolabial fold looks? at M11/2: Not satisfied | 27 | 26
  Are you satisfied with how your nasolabial fold looks? at M3: number analyzed (Participants) | 53 | 53
  Are you satisfied with how your nasolabial fold looks? at M3: Satisfied | 34 | 33
  Are you satisfied with how your nasolabial fold looks? at M3: Not satisfied | 19 | 20
  Are you satisfied with how your nasolabial fold looks? at M6: number analyzed (Participants) | 53 | 53
  Are you satisfied with how your nasolabial fold looks? at M6: Satisfied | 38 | 37
  Are you satisfied with how your nasolabial fold looks? at M6: Not satisfied | 15 | 16
  Are you satisfied with how your nasolabial fold looks? at M9: number analyzed (Participants) | 48 | 48
  Are you satisfied with how your nasolabial fold looks? at M9: Satisfied | 32 | 29
  Are you satisfied with how your nasolabial fold looks? at M9: Not satisfied | 16 | 19
  Are you satisfied with how your nasolabial fold looks? at M12: number analyzed (Participants) | 47 | 47
  Are you satisfied with how your nasolabial fold looks? at M12: Satisfied | 34 | 33
  Are you satisfied with how your nasolabial fold looks? at M12: Not satisfied | 13 | 14
  Are you satisfied with how your nasolabial fold looks? at M18: number analyzed (Participants) | 49 | 49
  Are you satisfied with how your nasolabial fold looks? at M18: Satisfied | 32 | 29
  Are you satisfied with how your nasolabial fold looks? at M18: Not satisfied | 17 | 20
  Are you satisfied with how your nasolabial fold looks? at M24: number analyzed (Participants) | 49 | 49
  Are you satisfied with how your nasolabial fold looks? at M24: Satisfied | 25 | 24
  Are you satisfied with how your nasolabial fold looks? at M24: Not satisfied | 24 | 25
  The result is aesthetically satisfying at M11/2: Satisfied | 29 | 28
  The result is aesthetically satisfying at M11/2: Not satisfied | 26 | 27
  The result is aesthetically satisfying at M3: number analyzed (Participants) | 52 | 51
  The result is aesthetically satisfying at M3: Satisfied | 31 | 30
  The result is aesthetically satisfying at M3: Not satisfied | 21 | 21
  The result is aesthetically satisfying at M6: number analyzed (Participants) | 53 | 53
  The result is aesthetically satisfying at M6: Satisfied | 37 | 36
  The result is aesthetically satisfying at M6: Not satisfied | 16 | 17
  The result is aesthetically satisfying at M9: number analyzed (Participants) | 48 | 48
  The result is aesthetically satisfying at M9: Satisfied | 31 | 29
  The result is aesthetically satisfying at M9: Not satisfied | 17 | 19
  The result is aesthetically satisfying at M12: number analyzed (Participants) | 47 | 47
  The result is aesthetically satisfying at M12: Satisfied | 36 | 34
  The result is aesthetically satisfying at M12: Not satisfied | 11 | 13
  The result is aesthetically satisfying at M18: number analyzed (Participants) | 49 | 49
  The result is aesthetically satisfying at M18: Satisfied | 32 | 30
  The result is aesthetically satisfying at M18: Not satisfied | 17 | 19
  The result is aesthetically satisfying at M24: number analyzed (Participants) | 49 | 49
  The result is aesthetically satisfying at M24: Satisfied | 28 | 27
  The result is aesthetically satisfying at M24: Not satisfied | 21 | 22
  The result is natural at M11/2: Satisfied | 37 | 37
  The result is natural at M11/2: Not satisfied | 18 | 18
  The result is natural at M3: number analyzed (Participants) | 53 | 53
  The result is natural at M3: Satisfied | 40 | 37
  The result is natural at M3: Not satisfied | 13 | 16
  The result is natural at M6: number analyzed (Participants) | 53 | 53
  The result is natural at M6: Satisfied | 41 | 40
  The result is natural at M6: Not satisfied | 12 | 13
  The result is natural at M9: number analyzed (Participants) | 48 | 48
  The result is natural at M9: Satisfied | 37 | 34
  The result is natural at M9: Not satisfied | 11 | 14
  The result is natural at M12: number analyzed (Participants) | 47 | 47
  The result is natural at M12: Satisfied | 37 | 36
  The result is natural at M12: Not satisfied | 10 | 11
  The result is natural at M18: number analyzed (Participants) | 49 | 49
  The result is natural at M18: Satisfied | 35 | 35
  The result is natural at M18: Not satisfied | 14 | 14
  The result is natural at M24: number analyzed (Participants) | 48 | 49
  The result is natural at M24: Satisfied | 32 | 30
  The result is natural at M24: Not satisfied | 16 | 19
  The facial volumes are restored at M11/2: Satisfied | 24 | 25
  The facial volumes are restored at M11/2: Not satisfied | 31 | 30
  The facial volumes are restored at M3: number analyzed (Participants) | 52 | 52
  The facial volumes are restored at M3: Satisfied | 30 | 30
  The facial volumes are restored at M3: Not satisfied | 22 | 22
  The facial volumes are restored at M6: number analyzed (Participants) | 53 | 53
  The facial volumes are restored at M6: Satisfied | 31 | 34
  The facial volumes are restored at M6: Not satisfied | 22 | 19
  The facial volumes are restored at M9: number analyzed (Participants) | 48 | 48
  The facial volumes are restored at M9: Satisfied | 28 | 27
  The facial volumes are restored at M9: Not satisfied | 20 | 21
  The facial volumes are restored at M12: number analyzed (Participants) | 47 | 47
  The facial volumes are restored at M12: Satisfied | 30 | 28
  The facial volumes are restored at M12: Not satisfied | 17 | 19
  The facial volumes are restored at M18: number analyzed (Participants) | 49 | 49
  The facial volumes are restored at M18: Satisfied | 27 | 28
  The facial volumes are restored at M18: Not satisfied | 22 | 21
  The facial volumes are restored at M24: number analyzed (Participants) | 49 | 49
  The facial volumes are restored at M24: Satisfied | 22 | 21
  The facial volumes are restored at M24: Not satisfied | 27 | 28
  My features seem rested at M11/2: Satisfied | 26 | 27
  My features seem rested at M11/2: Not satisfied | 29 | 28
  My features seem rested at M3: number analyzed (Participants) | 53 | 53
  My features seem rested at M3: Satisfied | 32 | 32
  My features seem rested at M3: Not satisfied | 21 | 21
  My features seem rested at M6: number analyzed (Participants) | 53 | 53
  My features seem rested at M6: Satisfied | 35 | 35
  My features seem rested at M6: Not satisfied | 18 | 18
  My features seem rested at M9: number analyzed (Participants) | 47 | 48
  My features seem rested at M9: Satisfied | 31 | 29
  My features seem rested at M9: Not satisfied | 16 | 19
  My features seem rested at M12: number analyzed (Participants) | 47 | 47
  My features seem rested at M12: Satisfied | 32 | 30
  My features seem rested at M12: Not satisfied | 15 | 17
  My features seem rested at M18: number analyzed (Participants) | 48 | 49
  My features seem rested at M18: Satisfied | 28 | 29
  My features seem rested at M18: Not satisfied | 20 | 20
  My features seem rested at M24: number analyzed (Participants) | 49 | 49
  My features seem rested at M24: Satisfied | 25 | 25
  My features seem rested at M24: Not satisfied | 24 | 24

8. Secondary Outcome: Injector Satisfaction
Description: Percentage of participants
Time Frame: After initial injection (Day 0) and touch-up if applicable (Month 1^1/2)
Population: Intent To Treat population - any subject included and randomized in the study with at least a post-basal value
Measure: Count of Participants; unit: Participants
Arm/Group | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55
Participants
  Ease of injection after initial injection: Very satisfied | 32 | 29
  Ease of injection after initial injection: Satisfied | 18 | 21
  Ease of injection after initial injection: Somewhat satisfied | 5 | 5
  Ease of injection after initial injection: Somewhat dissatisfied | 0 | 0
  Ease of injection after initial injection: Dissatisfied | 0 | 0
  Ease of injection after initial injection: Very dissatisfied | 0 | 0
  Ease of injection after touch-up: number analyzed (Participants) | 52 | 52
  Ease of injection after touch-up: Very satisfied | 31 | 31
  Ease of injection after touch-up: Satisfied | 15 | 13
  Ease of injection after touch-up: Somewhat satisfied | 3 | 2
  Ease of injection after touch-up: Somewhat dissatisfied | 3 | 6
  Ease of injection after touch-up: Dissatisfied | 0 | 0
  Ease of injection after touch-up: Very dissatisfied | 0 | 0
  Mouldability after initial injection: Very satisfied | 35 | 34
  Mouldability after initial injection: Satisfied | 20 | 19
  Mouldability after initial injection: Somewhat satisfied | 0 | 1
  Mouldability after initial injection: Somewhat dissatisfied | 0 | 1
  Mouldability after initial injection: Dissatisfied | 0 | 0
  Mouldability after initial injection: Very dissatisfied | 0 | 0
  Mouldability after touch-up: number analyzed (Participants) | 52 | 52
  Mouldability after touch-up: Very satisfied | 29 | 29
  Mouldability after touch-up: Satisfied | 17 | 22
  Mouldability after touch-up: Somewhat satisfied | 6 | 1
  Mouldability after touch-up: Somewhat dissatisfied | 0 | 0
  Mouldability after touch-up: Dissatisfied | 0 | 0
  Mouldability after touch-up: Very dissatisfied | 0 | 0
  Ease of product positioning after initial injection: Very satisfied | 27 | 26
  Ease of product positioning after initial injection: Satisfied | 23 | 25
  Ease of product positioning after initial injection: Somewhat satisfied | 5 | 4
  Ease of product positioning after initial injection: Somewhat dissatisfied | 0 | 0
  Ease of product positioning after initial injection: Dissatisfied | 0 | 0
  Ease of product positioning after initial injection: Very dissatisfied | 0 | 0
  Ease of product positioning after touch-up: number analyzed (Participants) | 52 | 52
  Ease of product positioning after touch-up: Very satisfied | 26 | 25
  Ease of product positioning after touch-up: Satisfied | 23 | 25
  Ease of product positioning after touch-up: Somewhat satisfied | 2 | 2
  Ease of product positioning after touch-up: Somewhat dissatisfied | 1 | 0
  Ease of product positioning after touch-up: Dissatisfied | 0 | 0
  Ease of product positioning after touch-up: Very dissatisfied | 0 | 0
  Immediate result after initial injection: Very satisfied | 16 | 8
  Immediate result after initial injection: Satisfied | 31 | 32
  Immediate result after initial injection: Somewhat satisfied | 7 | 11
  Immediate result after initial injection: Somewhat dissatisfied | 1 | 4
  Immediate result after initial injection: Dissatisfied | 0 | 0
  Immediate result after initial injection: Very dissatisfied | 0 | 0
  Immediate result after touch-up: number analyzed (Participants) | 52 | 52
  Immediate result after touch-up: Very satisfied | 27 | 25
  Immediate result after touch-up: Satisfied | 24 | 25
  Immediate result after touch-up: Somewhat satisfied | 1 | 2
  Immediate result after touch-up: Somewhat dissatisfied | 0 | 0
  Immediate result after touch-up: Dissatisfied | 0 | 0
  Immediate result after touch-up: Very dissatisfied | 0 | 0
  Result after massage (initial inejction): Very satisfied | 15 | 10
  Result after massage (initial inejction): Satisfied | 31 | 33
  Result after massage (initial inejction): Somewhat satisfied | 8 | 9
  Result after massage (initial inejction): Somewhat dissatisfied | 1 | 3
  Result after massage (initial inejction): Dissatisfied | 0 | 0
  Result after massage (initial inejction): Very dissatisfied | 0 | 0
  Result after massage (touch-up): number analyzed (Participants) | 52 | 52
  Result after massage (touch-up): Very satisfied | 26 | 26
  Result after massage (touch-up): Satisfied | 26 | 26
  Result after massage (touch-up): Somewhat satisfied | 0 | 0
  Result after massage (touch-up): Somewhat dissatisfied | 0 | 0
  Result after massage (touch-up): Dissatisfied | 0 | 0
  Result after massage (touch-up): Very dissatisfied | 0 | 0

9. Secondary Outcome: Collection of Injection Site Reactions
Description: Proportion of subjects presenting at least one ISR of any severity
Time Frame: Day 0, Month 1^1/2, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
Population: Safety population - any subject having used the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55
Participants
  D0 after initial injection: No sign | 3 | 6
  D0 after initial injection: At least one sign | 52 | 49
  M11/2 before touch-up: No sign | 50 | 54
  M11/2 before touch-up: At least one sign | 5 | 1
  M11/2 after touch-up: number analyzed (Participants) | 52 | 52
  M11/2 after touch-up: No sign | 1 | 5
  M11/2 after touch-up: At least one sign | 51 | 47
  M3: number analyzed (Participants) | 49 | 49
  M3: No sign | 44 | 47
  M3: At least one sign | 5 | 2
  M6: number analyzed (Participants) | 53 | 53
  M6: No sign | 49 | 51
  M6: At least one sign | 4 | 2
  M9: number analyzed (Participants) | 48 | 48
  M9: No sign | 45 | 46
  M9: At least one sign | 3 | 2
  M12: number analyzed (Participants) | 47 | 47
  M12: No sign | 43 | 45
  M12: At least one sign | 4 | 2
  M18: number analyzed (Participants) | 49 | 49
  M18: No sign | 47 | 48
  M18: At least one sign | 2 | 1
  M24: number analyzed (Participants) | 49 | 49
  M24: No sign | 47 | 49
  M24: At least one sign | 2 | 0

10. Secondary Outcome: Collection of Adverse Events
Description: Number of Adverse Events (AEs) Number of Adverse Device Effects (ADEs) Proportion of subjects with at least one AE Proportion of subject with at least one ADE
Time Frame: Day 0 to Month 24
Population: Safety population - any subject having used the investigational device
Measure: Number; unit: participants
Units Other Than Participants: Nasolabial fold
Groups:
- Gana V: Participants received Gana V in one nasolabial fold (as per randomization list-split face design).
- Sculptra: Participants received Sculptra in one nasolabial fold (as per randomization list-split face design).
Arm/Group | Gana V Versus Sculptra | Gana V | Sculptra
Number analyzed (Participants) | 55 | 55 | 55
Number analyzed (Nasolabial fold) | 110 | 55 | 55
participants
  Proportion of subjects with at least one AE : With | 43 | 43 | 43
  Proportion of subjects with at least one AE : Without | 12 | 12 | 12
  Proportion of subjects with at least one SAE : With | 1 | 1 | 1
  Proportion of subjects with at least one SAE : Without | 54 | 54 | 54
  Proportion of subjects with at least one ADE : With | 18 | 17 | 14
  Proportion of subjects with at least one ADE : Without | 37 | 38 | 41
  proportion of subects with at least one SADE : With | 0 | 0 | 0
  proportion of subects with at least one SADE : Without | 55 | 55 | 55

ADVERSE EVENTS:
Time Frame: 24 months
Description: Definitions from MDCG were used as the study was done on a medical device
Arm/Group | Gana V | Sculptra
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55 | 1/55
Other Adverse Events (participants affected / at risk) | 42/55 | 42/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gana V (N=55) | Sculptra (N=55)
Femoral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gana V (N=55) | Sculptra (N=55)
Eye disorder (Eye disorders) | 2 (2) | 2 (2) — Glaucoma / conjunctivitis
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (6) | 5 (6) — Gastroenteritis, bloating, reflux
General disorders and administration site conditions (General disorders) | 29 (70) | 30 (64)
Infection (Infections and infestations) | 15 (19) | 15 (19)
Muskulokeletal disorders (Musculoskeletal and connective tissue disorders) | 11 (17) | 11 (17)
Headache / Migraine (Nervous system disorders) | 14 (50) | 14 (50)
Pneumonia / Tracheitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Acne, seborrheic dermatitis, burn (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
* Primary assessment subjective
* Low quantity of product injected compared to other study found in the litterature
* Comparator chosen is not the same concentration as Gana V

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT05215054/Prot_SAP_000.pdf